CLINICAL TRIAL: NCT02132871
Title: Noninvasive Assessment of Preload Dependency by Passive Leg Raising Test and Impedance Cardiography Compared to Echocardiographic Measurements After Cardiac Surgery
Brief Title: Preload Dependency by Impedance Cardiography After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5516
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Cardiac Surgery With Extracorporeal Circulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Device: Impedance cardiography Physioflow ®

INTERVENTIONS:
Device: Impedance cardiography Physioflow ®

SUMMARY:
The primary purpose of this study is to investigate wether the measure of stroke volume (SV) variations by impedance cardiography during passive leg raising (PLR) can reliably predict preload dependency after cardiac surgery, in comparison to a reference parameter : velocity time integral (VTI) variation measured by transthoracical echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Men or women over 18 years
* Affiliated to a social protection
* Signed written consent
* Informed about the results of the medical visit
* All type of cardiac surgery with extracorporeal circulation performed at University Hospital of Strasbourg
* Sedated and under mechanical ventilation

Exclusion Criteria:

* Cardiac arrhythmia
* Contraindication to PLR maneuver
* Exclusion period due to inclusion in a previous or ongoing study
* Impossibility to provide enlightened information
* Patient deprived of liberty, under judicial protection, trusteeship or guardianship
* Pregnancy, lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Area under ROC curve comparing SV variation (impedance cardiography) and VTI variation after PLR | Within the 6 first hours after cardiac surgery
  Patients classified as responders and non responders to PLR : VTI variation ≥ 12% or < 12%

SECONDARY OUTCOMES:
Variation of central veinous pressure, left auricular pressure and left ventricular filling pressures after PLR (ROC curves, correlation tests) | Within the 6 first hours after cardiac surgery
Respiratory variation of inferior vena cava | Within the 6 first hours after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nassim HESHMATI, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service d'Anesthésiologie, Nouvel Hôpital Civil, Hôpitaux Universitaires de Strasbourg, Strasbourg, France